CLINICAL TRIAL: NCT00939497
Title: Bioequivalence Study of Risperidone 1.0 mg Tablets of Torrent Pharmaceuticals Limited., India and Risperdal® (Risperidone) 1.0 mg Tablets of Janssen Pharmaceutical Products, LP, USA, in Healthy Human Adult Subjects, Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Other Study IDs: 1119/07
Record Dates: First submitted 2009-07-10; First posted 2009-07-15 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Healthy
MeSH Terms: interventions — Risperidone

INTERVENTIONS:
Drug: Risperidone

SUMMARY:
Objective:

* To assess the bioequivalence of Risperidone 1.0 mg tablets of Torrent Pharmaceuticals Limited., India and Risperdal® (Risperidone) 1.0 mg tablets of Janssen Pharmaceutical Products, LP, USA, in healthy human adult subjects, under fasting conditions.

Study Design:

* A randomized, open label, two treatment, two period, two sequence, single dose, crossover study, under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy human adult subjects between 18-55 years of age (inclusive), having a body mass index (BMI) between 18 and 27 kg/m2.
2. Subjects who have no evidence of underlying disease during screening history and whose physical examination is performed within 21 days prior to commencement of the study.
3. Subjects whose screening laboratory values are within normal limits or considered by the physician/Principal Investigator to be of no clinical significance.
4. Informed consent given in written form according to section 11.3 of the protocol.
5. Female Subjects:

   * Of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence.
   * Postmenopausal for at least 1 year.
   * Surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject).

Exclusion Criteria:

1. History or presence of significant:

   * Cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, musculoskeletal, neurological or psychiatric disease.
   * Alcohol dependence, alcohol abuse or drug abuse within past one year.
   * Moderate to heavy smoking (>10 cigarettes/day) or consumption of tobacco products.
   * History of difficulty in swallowing tablet / capsule.
   * Clinically significant illness within 4 weeks before the start of the study
   * Asthma, urticaria or other allergic type reactions after taking any medication.
   * Positive urine drug screening, HIV, Hepatitis B & C tests.
   * Any history of hypersensitivity to Risperidone.
   * Existence of any surgical or medical condition, which, in the judgment of clinical investigator might interfere with the pharmacokinetics of the drug or likely to compromise the safety of the subject.
   * Inability to communicate or co-operate with the investigator due to language problem, attitude, poor mental development / impaired cerebral function.
2. Subject who has participated in any other clinical trial involving drug administration and collection of blood samples or has donated blood in the preceding 12 weeks prior to the start of the study.
3. Subjects who have:

   * Systolic blood pressure less than 90 mm of Hg or more than 150 mm of Hg.
   * Diastolic blood pressure less than 60 mm of Hg or more than 94 mm of Hg. Minor deviations (2-4 mm Hg) at check-in may be acceptable at the discretion of the physician /investigator.
   * Pulse rate below 50/minute or above 105/minute.

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- Lotus Labs Pvt. Ltd., Bangalore, Karnataka, India